CLINICAL TRIAL: NCT01506973
Title: A Phase I/II/Pharmacodynamic Study of Hydroxychloroquine in Combination With Gemcitabine/Abraxane to Inhibit Autophagy in Pancreatic Cancer
Brief Title: A Study of Hydroxychloroquine in Combination With Gemcitabine/Abraxane in Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19211
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Advanced Adenocarcinoma; Metastatic Adenocarcinoma
Keywords: histologically or cytologically documented
MeSH Terms: conditions — Adenocarcinoma | interventions — Hydroxychloroquine; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine/Abraxane/Hydroxychloroquine (Experimental): Abraxane: 125mg/m2 IV infusion over 30 minutes on Days 1, 8, 15 Gemcitabine: 1000mg/m2 IV infusion over 30-100 minutes on Days 1, 8, 15 Hydroxychloroquine: 1200 mg/day PO daily (600mg BID) Daily from D1
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gemcitabine; Drug: Abraxane
- Gemcitabine/Abraxane (Experimental): Abraxane: 125mg/m2 IV infusion over 30 minutes on Days 1, 8, 15 Gemcitabine: 1000mg/m2 IV infusion over 30-100 minutes on Days 1, 8, 15
  Interventions: Drug: Gemcitabine; Drug: Abraxane

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — no other names
  Arms: Gemcitabine/Abraxane/Hydroxychloroquine
Drug: Gemcitabine — no other names
Drug: Abraxane — no other names

SUMMARY:
In this Phase I/II clinical trial, the investigators seek to pilot the addition of Hydroxychloroquine (HCQ) to a commonly-used front-line therapy of pancreatic cancer, gemcitabine/nab-paclitaxel. The investigators plan a run-in to define tolerable doses, and will explore doses of 800 and 1200 mg/day in successive cohorts of 6 patients. The investigators will assess toxicity continuously, and determine the dose for the Phase II trial based on standard toxicity criteria.

The correlative endpoints of this trial are directed to the pharmacokinetics of HCQ, and pharmacokinetic model of HCQ based on data from several ongoing trials, and the data from these patients will contribute to refining the model. The investigators will analyze both measured and model-predicted indices for their relationship to autophagy induction. Autophagy will be assessed as the accumulation of autophagocytic vesicles in the PMNs of treated patients, together with the induction of the expression of autophagy-related proteins on western analysis, quantitated by densitometry. The investigators will document the rates of metabolic response as a consequence of treatment, as a therapeutic marker that may be related to the degree of autophagy inhibition. Since the investigators have previously demonstrated a key role of JNK1 in the induction of autophagy by chemotherapy, the investigators will analyze archival tumor materials to determine variability in this marker, as a baseline for potential future trials. Finally, this study will incorporate metabolic profiling by mass spectrometry, which will be related to mutations (including Kras) in pretreatment tumor specimens. Mutational analysis will be accomplished by targeted sequencing or by next-generation sequencing, and the need for fresh tissue for all these endpoints will require patients to have a biopsy performed before treatment at at 6-8 weeks after beginning treatment. In the previous study of the Hh inhibitor GDC-0973 with the same chemotherapy, the investigators were able to obtain repeat biopsies successfully on all patients. The importance of these biopsies, to move the science forward in an era in which the tools now exist to provide meaningful correlative science, cannot be overstated.

DETAILED DESCRIPTION:
Recent strategies have focused on improving the efficacy of gemcitabine either by improving the method of delivery, or by combining gemcitabine with other non-cross resistant agents. A sequence of Phase III combination studies of gemcitabine in combination (with oxaliplatin, and with the targeted therapies bevacizumab and cetuximab) have been negative, though based on strikingly positive Phase II data generated in cancer centers. Several studies suggest that taxanes are active in pancreatic cancer, but a randomized trial of gemcitabine with taxanes has not been preformed, probably on the basis that the differences in Phase II were insufficiently persuasive. The development of a novel taxane conjugate with albumin, abraxane, with established activity in breast cancer, prompted a Phase II trial of gemcitabine/abraxane by Von Hoff (6). Phase I/II data were highly promising, with response rates of the order of 40%, with tolerable toxicity, and a one-year survival of about 48%. A phase III trial of gemcitabine versus gemcitabine/abraxane is in progress, and based on these promising data has served as the control chemotherapy for previous SU2C trials. The development of a more intensive, but toxic regimen (FOLFIRINOX) in no way diminishes the enthusiasm for this chemotherapy backbone, given the activity in Phase II trials that appears comparable (7). Given the promise of this regimen, and the possibility of making a substantial improvement in outcome with additional targeted interventions, we propose to continue to use this regimen in the current study.

Of particular interest in extending these studies to pancreatic cancer is the finding that autophagy inhibition is particularly deleterious to cell lines bearing a mutant Kras protein. Additional studies as part of the SU2C pancreatic cancer project reveal that an autophagy program is activated in the presence of mutant Kras, and thus prompts the testing of this strategy in a setting in which Kras is commonly (about 85%) mutated (SU2C, unpublished data).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented advanced or metastatic adenocarcinoma of the pancreas.
* Patients must have measurable disease as defined by the RECIST criteria as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20mm with conventional techniques on either CT or MRI. Marker (CA19-9 or CEA) elevation alone is insufficient for entry.
* Patients may have had prior adjuvant treatment for pancreatic cancer. The last dose of chemotherapy must have been 4 months prior to study entry.
* Patients with prior radiotherapy are acceptable. It must be at least 4 months since administration of radiation therapy and all signs of toxicity must have abated.
* Patients must be age 18 years or older.
* Patients must have an ECOG performance status of 0-1.
* The following required Initial Laboratory Values should be obtained within 4 weeks of the start of treatment:

  * Granulocytes 1,500/ml
  * Platelet Count 100,000/ml
  * Creatinine 1.5 x upper limit of normal
  * Bilirubin 1.5 x upper limit of normal
  * AST 5 x upper limit of normal
* Patients must not be pregnant or lactating as chemotherapy is thought to present substantial risk to the fetus/infant.
* Patients must have an accessible primary tumor or metastasis, and be willing to have a pre-treatment and post-treatment tumor biopsy (at 6 to 8 weeks after beginning).
* Patients must have a life expectancy of greater than three months.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Known allergy to HCQ
* Patients with previous treatment with abraxane.
* Patients on therapeutic doses of Coumadin ( 1 mg daily). The use of therapeutic or prophylactic low molecular weight heparin or fragmin is permitted.
* Patients with known G6PD deficiency, severe psoriasis, porphyria, macular degeneration or severe diabetic retinopathy are ineligible because of the potential for greater HCQ toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-12; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Karasic TB, O'Hara MH, Loaiza-Bonilla A, Reiss KA, Teitelbaum UR, Borazanci E, De Jesus-Acosta A, Redlinger C, Burrell JA, Laheru DA, Von Hoff DD, Amaravadi RK, Drebin JA, O'Dwyer PJ. Effect of Gemcitabine and nab-Paclitaxel With or Without Hydroxychloroquine on Patients With Advanced Pancreatic Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):993-998. doi: 10.1001/jamaoncol.2019.0684. PMID 31120501